CLINICAL TRIAL: NCT03640260
Title: Effects of Respiratory Regulation With Biofeedback in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Respiratory Regulation With Biofeedback in COPD
Acronym: RRBCOPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, I Ting Hsiao, Registered Nurse, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 180501
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): The experiment arm will get educational leaflets to pursed-lip with diaphragmatic breathing training and oximetry level evaluation.
  Interventions: Behavioral: breathing regulation with physical activity
- controlled (No Intervention)

INTERVENTIONS:
Behavioral: breathing regulation with physical activity — The subjects will have education leaflets with breathing and oximetry level evaluation training.
  Arms: experimental

SUMMARY:
Dyspnea is the main reason that patient with chronic obstructive pulmonary disease(COPD) to sedentary. It's a vicious circle of deteriorating lung function. The heart rate various(HRV)biofeedback with respiratory regulation training had been reported to reduce dyspnea and improve regulatory physical activities in COPD. However, HRV is not available with patients in communities persistently, the arm of this study is to explore the effect of the pulse oximeter biofeedback with respiratory regulation training to improve physical activities in COPD. A 2-group, randomized design study, the subjects are GOLD stage II-IV COPD from a medical center hospital of the middle of Taiwan. The experiment cases will be taught the skills of evaluating oximeter data and performing correct pursed-lip with diaphragmatic breathing. All experiment and controlled patients have to fill out the demographic form, the modified British Medical Research Council (mMRC), the international physical Activity questionnaire- short form(IPAQ-SF), exercise self-regulation efficacy scale (Ex-SRES), COPD assessment test (CAT), and physical activity & respiratory training diary in pre-intervention and 12 weeks later. The collective data will analyze with SPSS 22.0.

DETAILED DESCRIPTION:
Before subjects begin participation in any study-specific procedures, the investigators get institutional review board approval of the protocol, informed consent form, questionnaires and all subject information. A subject is considered enrolled when the investigator decides that the subject has met all eligibility criteria. All subjects must personally sign and date the IRB approved ICF before commencement of study-specific procedures. Each subject who enters the screening period for the study will receive a unique subject identification number before any study-related activities are performed. This number will be used to identify the subject throughout the study.

116 subjects will spend 20~30 minutes to fill out based demographic forms, mMRC, CAT, IPAQ, Ex-SRES and simple emotion questionnaires, then be randomized by sealed envelope to 1 of 2 arms. Under routine care, the experiment arm will get educational leaflets to pursed-lip with diaphragmatic breathing training and oximetry level evaluation. The controlled arm also has education leaflets but without breathing and oximetry level evaluation training. They be required to record respiratory regulation and physical activity diary while home care period up to first following out-patient department (about 12 weeks later). In the home care period, there are three times phone monitors to remind keep recording diary at first, forth and eighth week. Finally, mMRC, CAT, IPAQ and Ex-SRES will be finished again when first follow visit.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed COPD, pulmonary spirometry test FEV1/FVC<70% and FEV1<80%.
* 2. At least 20 years old and has communicative capacity.
* 3. Can walk by self or assistive device prior hospitalization.

Exclusion Criteria:

* 1. acute exacerbation attack or recurrent acute exacerbation and SpO2< 90%.
* 2. Can perform respiratory regulation correctly within exercising regularly.
* 3. Know cancer.
* 4. Comorbidity with sever pulmonary and cardiac disease.
* 5. Diseases of musculoskeletal system.
* 6. Psychotic or cognitive disorder that likely not be available to complete study procedures.
* 7. the hearing-impaired or visually disabled.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
adherence - evaluated by diary record | 12 weeks
  adherence of breathing and physical activity will be evaluated by diary record

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Changhua County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided